CLINICAL TRIAL: NCT04700319
Title: CAR-T CD19/CD20 for Patients With Advanced CD19/CD20+ B Cell Line Recurrent or Refractory Hematological Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PA-CART-1920-I -001
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: CAR
Keywords: B cell line; hematological malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD20 CAR-T cell infusion (Experimental): CD19/CD20 CAR-T cell infusion on relapsed or refractory hematological malignancies of CD19 / CD20+ B cell line
  Interventions: Drug: CD19/CD20 CAR-T cell infusion

INTERVENTIONS:
Drug: CD19/CD20 CAR-T cell infusion — CD19/CD20 CAR-T,Infusion,iv,0.2×10^6-5×10^6γδT /kg,once
  Other Names: Targeting CD19、CD20 autologous chimeric antigen receptor T cells#

SUMMARY:
This is a clinical study of CD19 / CD20 CAR-T cell infusion in the treatment of relapsed or refractory hematological malignancies in CD19 / CD20 positive B cell lines.

The aim of this study was to evaluate the efficacy and safety of autologous chimeric antigen receptor T cell infusion targeting CD19/CD20 in the treatment of relapsed or refractory CD19 / CD20 positive B cell line hematological malignancies.

DETAILED DESCRIPTION:
CD19 and CD20 are two proteins expressed in normal B cells and various B cell-derived hematological malignancies, including non Hodgkin's lymphoma (NHL), acute lymphoblastic leukemia (all) and chronic lymphoblastic leukemia (CLL). CD19 and CD20 are restricted to the surface of B cells. They are not expressed in hematopoietic stem cells, nor in other tissue cells. They exist in all stages of B cell development and differentiation. They are not lost from the cell surface until B cells differentiate into plasma cells. Clinical studies have found that CD19 and CD20 are excellent targets for immunotherapy of B-cell malignancies.The purpose of this study was to observe the efficacy and safety of treatment for patients with relapsed or refractory CD19 / CD20 positive B cell line hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

Only subjects meeting all of the following conditions were included in the study:

* The subjects who voluntarily participated in the study and signed the written informed consent;
* The age at the time of signing the informed consent is 3-70 years old, regardless of gender or race;
* The patients with CD19 / CD20 positive hematological malignancies without other effective treatment options include those who are not suitable for allogeneic stem cell transplantation (SCT) due to the following reasons:Age; Concurrent diseases; Other contraindications, such as total body irradiation (TBI) contraindications (TBI is one of the important treatment measures before allogeneic stem cell transplantation in all patients); Lack of suitable donors;
* Expected survival > 12 weeks;
* Relapse after any stem cell transplantation (no matter what previous treatment plan); and;
* Patients who relapsed after previous allogeneic SCT (myeloablative or non myeloablative) and met all other inclusion criteria:

  1. There was no active GVHD and no immunosuppression was required;
  2. Transplantation lasted more than 4 months;
* Serum creatinine ≤ 1.6 mg / dl and / or urea nitrogen ≤ 1.5 mg / dl;
* Serum AST and alt ≤ 5 x upper limit of normal value (ULN);
* It is necessary to have indicators for disease detection or evaluation, including detection of minimal residual disease (MRD) by immunophenotyping, cytogenetics or PCR;
* Cardiac function: left ventricular ejection fraction greater than or equal to 40%;
* ECoG physical condition (PS) ≤ 2;
* The pregnant test results of fertile female subjects within 48 hours before the infusion were negative and they were not in lactation period; all fertile female subjects took adequate contraceptive measures before entering the study and within 3 months after stopping the last infusion during the whole study period.

Exclusion criteria:

* Pregnant or lactating female patients;
* Participate in another clinical trial within 4 weeks before the study, or intend to participate in another clinical trial during the whole study period;
* Uncontrolled active infection;
* The history of human immunodeficiency virus is known;
* Active hepatitis B or hepatitis C infection;
* The systemic steroid treatment is needed during cell infusion or cell collection, or there are some diseases that researchers think may need steroid treatment during blood collection or infusion. In addition to cell collection or infusion, steroids for disease treatment are allowed, and inhaled steroids or hydrocortisone for physiological replacement therapy in patients with adrenocortical insufficiency are also allowed;
* There are grade 2-4 acute or systemic chronic GVHD;
* There is GVHD under treatment;
* Patients with cns3 disease progression or central nervous system parenchymal lesions that may increase central nervous system toxicity; patients with active central nervous system leukemia or lymphoma infiltration;
* Absolute neutrophil count < 750 / μ L or platelet count < 50000 / μ l caused by non primary diseases;
* When collecting cells, they received systemic chemotherapy 2 weeks ago or radiotherapy 3 weeks ago;
* Researchers believe that it is not suitable to participate in this clinical trial due to various reasons.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR 3 | three months after CAR-T cells infusion
  3-month objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, Principal Investigator — No.1, Swan Lake Road, new administrative and Cultural District, Hefei City, Anhui Province
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China